CLINICAL TRIAL: NCT02945475
Title: Neural Mechanisms for Appetitive Responses to High Reward Foods
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Kathleen Page, Associate Professor of Medicine, University of Southern California
Other Study IDs: HS-09-00395
Record Dates: First submitted 2016-06-28; First posted 2016-10-26 (Estimated); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Appetitive Behavior; Obesity
Keywords: functional magnetic resonance imaging; eating behavior; sugar
MeSH Terms: conditions — Appetitive Behavior; Obesity; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- obese: Individuals ages 18 to 35 years of age with body mass index (BMI) 30-40 kg/m2
- lean: Individuals ages 18 to 35 years of age with BMI of 19-24.9 kg/m2
- overweight: Individuals ages 18 to 35 years of age with BMI of 25-29.9 kg/m2

SUMMARY:
This study is aimed at understanding neuroendocrine responses to different types of sugars and how this influences feeding behavior among lean, overweight, and obese individuals.

DETAILED DESCRIPTION:
The investigators have previously combined functional magnetic resonance imaging (fMRI) with hormonal and behavioral assessments to better understand the impacts of glucose and fructose on appetite and its central regulation in humans and have made important observations in lean individuals linking fructose consumption to overeating and obesity. The investigators now propose to expand this work by examining the impacts of glucose and fructose ingested together (sucrose), as occurs in real life, and by examining effects of a common non-nutritive sweetener, sucralose, on brain and appetitive response. The investigators propose a random-order crossover design to determine the effects of caloric and non-nutritive sweeteners among lean, overweight, and obese participants. The investigators will measure circulating levels of hormones involved in satiety signaling, quantify food intake, and measure brain activity using blood-oxygen level dependent and arterial spin labeling methods and functional connectivity analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years, right-handed, weight change <2% for at least 3 months prior to participation, no history of diabetes or other significant medical problems, fasting glucose <126 mg/dl.
* Lean group: BMI of 19-24.9 kg/m2
* Obese Group: BMI 30-40 kg/m2
* Overweight Group: BMI of 25-29.9 kg/m2

Exclusion Criteria:

* Neurological, psychiatric or addiction disorder, fasting glucose ≥126 mg/dl, use of prescription medication (with the exception of contraceptives), tobacco use, contraindications to MRI scanning (detailed in Protection of Human Subjects), fructose intolerance, history of eating disorder, actively trying to lose weight.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants in the greater Los Angeles area will be recruited. Lean, overweight, and obese participants will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2016-02; Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Changes of Blood oxygen level-dependent (BOLD) signal responses to food vs non-food cues after ingestion of different types of sugar. BOLD signal responses to food cues will be compared at the level of whole brain and within a priori regions of interest. | Sessions 1, 2, 3, 4
  These will be compared between ingestion of drinks and at level of whole brain and in regions of interest
Cerebral Blood Flow Response | Sessions 1, 2, 3, 4
  Arterial spin labeling with be used to determine brain areas with relative increases or decreases in CBF after ingestion of sucrose, glucose, or sucralose.
Systemic Metabolite and Hormone Responses | Sessions 1, 2, 3, 4
  The effects of sugar ingestion on changes in systemic metabolite (glucose) and hormone (insulin, GLP-1, leptin, ghrelin, peptide YY) levels will be assessed.

SECONDARY OUTCOMES:
Functional Connectivity between regions involved in regulation of food intake | Sessions 1, 2, 3, 4
  Investigators will perform a physiological-psychological-interaction (PPI) analysis using the nucleus accumbens as the seed to explore brain regions showing increased functional connectivity to the seed during the food-cue task.
Appetite Ratings | Sessions 1, 2, 3, 4
  Ratings of hunger and desire for food in response to food vs non-food cues will be analyzed using a repeated-measures ANOVA with condition (glucose, sucrose, sucralose) and stimulus (food vs non-food) as within-subject factors.
Ad Libitum Food Intake | Sessions 1, 2, 3, 4
  Total calories consumed and percent calories from sugar, fat and protein will be compared between conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Page, MD, Principal Investigator — University of Southern California
Locations (1):
- Alexandra Yunker, Los Angeles, California, United States

REFERENCES:
- [Derived] Chakravartti SP, Jann K, Veit R, Liu H, Yunker AG, Angelo B, Monterosso JR, Xiang AH, Kullmann S, Page KA. Non-caloric sweetener effects on brain appetite regulation in individuals across varying body weights. Nat Metab. 2025 Mar;7(3):574-585. doi: 10.1038/s42255-025-01227-8. Epub 2025 Mar 26. PMID 40140714
- [Derived] Smith A, Page KA, Smith KE. Associations between affect dynamics and eating regulation in daily life: a preliminary ecological momentary assessment study. Cogn Emot. 2024 Aug;38(5):818-824. doi: 10.1080/02699931.2024.2323478. Epub 2024 Mar 1. PMID 38427387
- [Derived] Alves JM, Yunker AG, Luo S, Jann K, Angelo B, DeFendis A, Pickering TA, Smith A, Monterosso JR, Page KA. FGF21 response to sucrose is associated with BMI and dorsal striatal signaling in humans. Obesity (Silver Spring). 2022 Jun;30(6):1239-1247. doi: 10.1002/oby.23432. Epub 2022 May 2. PMID 35491674
- [Derived] Yunker AG, Alves JM, Luo S, Angelo B, DeFendis A, Pickering TA, Monterosso JR, Page KA. Obesity and Sex-Related Associations With Differential Effects of Sucralose vs Sucrose on Appetite and Reward Processing: A Randomized Crossover Trial. JAMA Netw Open. 2021 Sep 1;4(9):e2126313. doi: 10.1001/jamanetworkopen.2021.26313. PMID 34581796
- [Derived] Yunker AG, Luo S, Jones S, Dorton HM, Alves JM, Angelo B, DeFendis A, Pickering TA, Monterosso JR, Page KA. Appetite-Regulating Hormones Are Reduced After Oral Sucrose vs Glucose: Influence of Obesity, Insulin Resistance, and Sex. J Clin Endocrinol Metab. 2021 Mar 8;106(3):654-664. doi: 10.1210/clinem/dgaa865. PMID 33300990